CLINICAL TRIAL: NCT05012969
Title: Investigation of Efficacy of Use of a Bandage to Prevent Hip Dislocation After Total Hip Arthroplasty in Patients With Previous Dislocation
Brief Title: Investigation of Efficacy of Use of a Bandage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HipStop
Record Dates: First submitted 2015-11-19; First posted 2021-08-19 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Hip Dislocation
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): HipStop bandage for 12 weeks to prevent dislocation of the hip
  Interventions: Device: Hipstop bandage
- control (No Intervention): normal procedure after dislocation of hip which is information on movement restrictions

INTERVENTIONS:
Device: Hipstop bandage — 12 weeks use of a bandage to prevent hip dislocations in patients with previous dislocations
  Arms: intervention

SUMMARY:
This trial investigates the effectiveness of using a bandage after dislocation of the hip after total hip arthroplasty.

Patients with a dislocated hip after total hip arthroplasty coming to the emergency department to have the hip relocated will be asked to participate in the trial. The patients will be randomised to either a bandage that reduces flexion, adduction and internal rotation of the hip or no bandage.

DETAILED DESCRIPTION:
This trial investigates the effectiveness of using a bandage after dislocation of the hip after total hip arthroplasty.

Patients with a dislocated hip after total hip arthroplasty coming to the emergency department to have the hip relocated will be asked to participate in the trial. The patients will be randomised to either a bandage that reduces flexion, adduction and internal rotation of the hip or no bandage. Patients in the intervention group will use the bandage for 12 weeks and patients in the control group will receive the normal treatment which is information by a physiotherapist on movement restrictions.

50 patients will be allocated in the intervention group and 50 patients will be allocated to the control group.

We will investigate:

1. Whether there is a difference in number of dislocations between the two groups in the project period (12 weeks).
2. Patients' hip function, quality of life and satisfaction with the treatment in the two groups
3. The safety, wear and durability of the bandage after 12 weeks of use

ELIGIBILITY:
Inclusion Criteria:

* Has had at least one previous hip dislocation after total hip arthroplasty

Exclusion Criteria:

* Dislocation in other directions than posterior/superior
* Loose prosthesis
* wounds in the area of skin that is in contact with the bandage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-11; Primary Completion 2021-12 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
number of dislocations | 12 weeks

SECONDARY OUTCOMES:
Hip function | 12 weeks
  Oxford Hip Score, scores running from 0 to 48 with 48 being the best outcome
Helat-related quality of life | 12 weeks
  SF-36, a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability
Patient satisfaction | 12 weeks
  questions to patients
Safety, wear and durability of bandage | 12 weeks
  Questionnaire to physiotherapists

CONTACTS AND LOCATIONS:
Overall Officials: Inger Mechlenburg, PhD, Principal Investigator — University of Aarhus; Maiken Stilling, PhD, Principal Investigator — University of Aarhus
Locations (2):
- Denmark (2):
  - Holstebro Regional Hospital, Holstebro
  - Viborg Regional Hospital, Viborg